CLINICAL TRIAL: NCT01320410
Title: Clinical Trial to Evaluate the Pharmacokinetics, Safety, and Tolerance of Single Dose Administration of a New Injectable Prolonged Release Formulation of Risperidone Using ISM® Technology in Healthy Volunteers
Brief Title: Pharmacokinetics, Safety, and Tolerance Study of Single Dose Administration of Risperidone ISM®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rovi Pharmaceuticals Laboratories (Industry)
Allocation: Non-Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: ROV-RISP-2009-01
Record Dates: First submitted 2011-03-17; First posted 2011-03-22 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2011-03

CONDITIONS: Healthy

INTERVENTIONS:
Drug: ISM®

SUMMARY:
The study will comprise two dosing periods in two different cohorts of healthy volunteers. The investigators will begin with a single dosage period I (1 injection of 25 mg of Risperidone for each subject); single dosage period II, different from the previous one (1 injection of 37.5 mg of Risperidone for each subject), in a second group of healthy volunteers different from the first group will not start until after a preliminary analysis has been made of the safety data and plasma concentration data are known for the formulation of prolonged release Risperidone using the ISM® technology.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers of both sexes with a minimum age of 18 years and a maximum age of 50 years.
2. Healthy female volunteers should have a negative pregnancy test and, if they are of childbearing age, should use at least 2 medically accepted contraceptive methods.
3. Each volunteer must be capable of understanding enough to complete all tests and exams required in the protocol.
4. Each volunteer must understand the nature of the study and sign an informed consent document.
5. Vital signs (systolic and diastolic blood pressure, heart rate, and temperature) and ECG record within the normal range.
6. The results of the laboratory tests (complete blood count and biochemistry) and ECG should fall within the normal reference ranges or show minor deviations that the investigator does not consider clinically relevant.
7. The investigator must consider the volunteers suitable candidates for prolonged release intramuscular administration.
8. Healthy volunteers must have a body mass index between 19 and 27 kg/m2, and weigh between 50 and 100 kg.
9. Healthy volunteers may not have known cardiovascular disease, orthostatic hypotension, seizures, a family history of prolonged QT interval, bradycardia, electrolyte disturbances (hypokalemia, hypomagnesemia), or hyperprolactinemia.

Exclusion Criteria:

1. Pregnant women, nursing women, and female volunteers who are not using effective contraceptive methods.
2. Previous history of alcohol, drug, or substance abuse during the month prior to the selection. Average daily alcohol consumption exceeding 2 units (20 g/d). Smokers of more than 5-10 cigarettes per day in the 3 months prior to the start of the study.
3. History of allergy, idiosyncrasy, hypersensitivity or severe adverse reactions to medications, or contraindications to treatment with Risperidone as recorded in the data sheet of the drug.
4. Positive serology for hepatitis B or C, or for HIV.
5. History or clinical evidence of cardiovascular disease, respiratory, renal, hepatic, endocrine, gastrointestinal, hematological, neurological, psychiatric, or other chronic diseases that may interfere with the objectives of the trial.
6. Major consumer of stimulating beverages (> 5 cups of coffee, tea, cola drinks, or similar per day).
7. Positive urine test for ethanol, cannabis, cocaine, amphetamines, benzodiazepines, or opiates.
8. Baseline platelet number below 100,000/mm3 or serum potassium> 5.5 mEq / L.
9. Having undergone surgery in the past 6 months.
10. Plasma prolactin values outside the reference range (40 mcIU/ml to 530 mcIU/ml).
11. Having participated in another clinical trial during the three months before the start of the study.
12. Having donated blood within 4 weeks before the start of the study.
13. Having taken medication regularly in the month prior to the start of the study or symptomatic medication in the week before the start of the study, except for oral contraceptives, vitamins, herbal remedies, or dietary supplements that, according to the Principal Investigator or co-workers designated by him/her, do not involve a risk for the subjects and do not interfere with the objectives of the study.
14. Taking ASA and/or NSAIDs within 10 days before the start of the trial until the end of the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

PRIMARY OUTCOMES:
The main objective of the study is to evaluate the pharmacokinetics, safety, and tolerability